CLINICAL TRIAL: NCT06842238
Title: Descriptive Study of the Initial Management of Young Children With Moderate Acute BRONCHiotitis With Home Hospitalisation
Acronym: BRONCHAD
Status: Recruiting | Type: Observational
Sponsor: Elsan (Other)
Collaborators: HAD privée de Poitiers (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024-A01404-43
Record Dates: First submitted 2025-02-07; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Bronchiolitis; Bronchiolitis Acute
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The occurrence of a first episode of acute bronchiolitis in an infant or young child (3 months-2 years) always represents a medical event that generates stress for parents and in some cases for the primary care physician when it is necessary to decide on the child's orientation for treatment. Each year, during the winter season, this pathology affects 30% of infants under two years old (480,000 annual cases in France), generates approximately 30,000 hospitalizations and exposes to an overall mortality risk of 0.08%.

According to the recommendations of the HAS (2019), moderate bronchiolitis does not require systematic hospitalization and can be managed in a Home Hospitalization (HAD) context.

When the child's examination data do not find signs of severity, the SpO2 measurement is greater than 92% and the family context allows for return home, HAD management is a reasonable option and represents an alternative to the classic scheme of assessing the level of severity by the emergency department and subsequent hospitalization if necessary. HAD management is carried out within the framework of a very structured "patient pathway", codified and supervised by the pediatric teams and doctors of this department. This patient pathway concerns children with a moderate form of bronchiolitis without oxygen requirements at the time of inclusion. This must be 48 hours from the onset of the child's respiratory clinical signs.

The main objective of this study is to describe the need for oxygen therapy for a young child with moderate acute bronchiolitis syndrome during home hospitalization (HAD) care.

ELIGIBILITY:
Inclusion Criteria:

* Any infant with moderate bronchiolitis according to the HAS definition (except for the SpO2 criterion which must be greater than or equal to 92% to avoid the patient being on oxygen therapy upon admission)
* Age > 2 months and ≤ 2 years
* Respiratory syndrome for 48 hours
* Infant with a first episode of bronchiolitis
* Referral of the general practitioner/treating pediatrician for home hospitalisation care
* Parents' agreement for the choice of home hospitalisation care
* Non-opposition or free and informed consent of both parents to the use of the child's health data

Exclusion Criteria:

* Patient not receiving health protection
* Comorbidities: congenital heart disease with shunt, chronic pulmonary pathology including bronchopulmonary dysplasia, neuromuscular pathology, immune deficiency, multiple disabilities Congenital heart disease
* Refusal of one or both parents for the proposed pathway
* Doubts about the parents' understanding of the nature of home hospitalisation care
* Severe bronchiolitis or with saturation < 92%

  * Moderate bronchiolitis but evolving for less than 48 hours
  * Cases of psychiatric pathologies or depressive syndrome diagnosed in the parents.

Ages: 2 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Babies between 2 months and 2 years old
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Oxygenotherapy | one month
  Need for oxygen therapy during home hospitalisation care

SECONDARY OUTCOMES:
Oxygen therapy assistance | up to one month
  Oxygen therapy assistance during home hospitalization care
Home hospitalization support | up to one month
  Duration of home hospitalization support
Hospitalization time | up to one month
  hospitalization during home hospitalization care
QUALIN questionnaire | day 1, day 7 and one month
  QUALIN questionnaire is a 34-item scale to assess an infant's quality of life.
Hospital Anxiety and Depression Scale questionnaire | day 1, day 7 and one month
  HADS questionnaire has 14 items between 0 and more than 11 points
Direct costs | day 1, day 7 and one month
  daily cost of home hospitalization without oxygen, daily cost of home hospitalization with oxygen, GHS bronchiolitis level 2

CONTACTS AND LOCATIONS:
Locations (1):
- Polyclinique de Poitiers - HAD, Poitiers, France